CLINICAL TRIAL: NCT06312605
Title: Patient Response and Recurrence Rate Following Adjunctive Intra-Mucosal or Topical Ascorbic Acid To Gingival Depigmentation Using Surgical Scalpel Technique: (Randomized Clinical and Histological Trial)
Brief Title: The Adjunctive Role of Vitamin C on Pigment Recurrence (Randomized Clinical and Histological Trial)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Osama Mohamed Hashem, Demonstrator at oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 230620
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gingival Pigmentation
Keywords: Gingival pigmentation /Pigment recurrence /Vitamin C

STUDY DESIGN:
Intervention Model Description: All participants receive surgical depigmentation then either vitamin C is applied following 2 regimens
Who Masked: Outcomes Assessor
Masking Description: Coding of the groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intramucosal vitamin C injection (Active Comparator): After surgical gingival depigmentation, injectable vitamin C (Redox C 500 mg) using insulin syringe(29 Gauge 1cc 0.33mm x 8mm 5/16 needle) is applied at gingival sites 0.1 ml for each point that should be 3 mm. The regimen is done once weekly for a month then once a month for additional 5 months.
  Interventions: Procedure: Injectable applied vitamin C
- (Vitamin C topical gel (Active Comparator): After surgical gingival depigmentation, patients in this group apply ascorbic acid containing gel prepared by Nawah Scientific Research Center. The micro emulsion was prepared by mixing tween 20 (4.66% w/w) as surfactant and isopropanol (2.3% w/w) as co-surfactant using magnetic stirring then diluted drop-wise with Vitamin C solution in water (10% w/w). The formed micro emulsion was then converted into gel using Poloxamer 407 (20% w/w) that was added at 4°C under continuous magnetic stirring
  Interventions: Procedure: Topical applied Vitamin C
- Control group (Placebo Comparator): Surgical gingival depigmentation is carried out for these patients
  Interventions: Procedure: Surgical depigmentation only

INTERVENTIONS:
Procedure: Injectable applied vitamin C — Surgical gingival depigmentation is done for all participants, after then they receive injectable vitamin C
  Arms: Intramucosal vitamin C injection
Procedure: Topical applied Vitamin C — Surgical gingival depigmentation is done for all participants, after then they are instructed to apply topical vitamin C
  Arms: (Vitamin C topical gel
Procedure: Surgical depigmentation only — Surgical gingival depigmentation only without any drug
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to determine the role of vitamin C on recurrence of gingival pigment after patients who are healthy and esthetically concerned with it received surgical removal of this pigment. The main question[s] it aims to answer are:

* Pigment recurrence after one year.
* Patient satisfaction and histological response of tissues.

Participants will be asked to come on regular follow up visits one group will receive vitamin C injection other will be asked to apply topical vitamin C on a specific regimen.

Researcher will compare the groups who received injectable vitamin C with those who topically applied it to see the effect of each.

DETAILED DESCRIPTION:
Esthetic dentistry is currently concerned with the pivotal role of the gingival tissue along with the teeth color, shape and position to achieve a harmonious attractive smile.

Physiological gingival hyperpigmentation is attributed to the increased activity of melanocytes rather than the increased number; consequently the gingiva in these individuals reveals increased density of melanophores. There are several pigments that contribute to physiological gingival hyper pigmentation, the main contributory pigment is melanin that is synthesized by melanocytes. Melanocytes form melanosomes granules from the amino acid tyrosine converting it into a molecule called dehydroxyphenylalanine (DOPA) through a hydroxylation process catalyzed by tryosinase enzyme.

Surgical and non-surgical approaches have been utilized to treat gingival hyperpigmentation. De-epithelizing of the target region is the main concept for most of the surgical interventions using different techniques as de-epithelizing using surgical blade or bur abrasion, cryosurgery and laser.

Among the minimal invasive non-surgical approaches of treating gingival hyperpigmentation was vitamin C that yielded promising results in the previous few years as proved in different clinical trials and have been recently documented in systemic review by .Vitamin C binds to melanin effectively once introduced into the tissues with a consequent deficient in calcium and copper affecting both melanin formation and transportation.

One of the main challenges after treating gingival hyperpigmentation is pigment recurrence. Different theories tried to explain the reasons for recurrence, some attributed it to the three dimensional shape of rete pegs, others attributed it to the migration theory and capability of cells to migrate from existing neighboring areas . Recurrence of pigment had shown to be inevitable occurring with nearly equal ranges in the previously illustrated techniques.

Sheel et al illustrated no recurrence of gingival pigmentation was observed after 9 months follow up with the topical application of vitamin C after surgical gingival depigmentation in a case report. This case report highlighted the ancillary role of vitamin C in decreasing the recurrence rate of gingival pigment after depigmentation.

According to the researcher knowledge, up to this time, there were no further studies investigating the long-term effect of using vitamin C to gain gingival color stability after depigmentation. This study was conducted to compare efficacy of vitamin C either locally injected or topically applied after surgical gingival depigmentation on recurrence of pigment and patient satisfaction over one-year follow up.

ELIGIBILITY:
Inclusion Criteria:

Both genders aged from 18-40. Systemically free patients from any disease as evidenced by the health questionnaire, using modified Cornell medical index and classified as ASA class I.

Patients who were diagnosed to have physiological gingival melanin pigmentation on the maxillary or mandibular keratinized gingiva with Dummett oral pigmentation score 2 or more.

Patients with thick gingival phenotype ≥ 1.5 mm.

Exclusion criteria:

Pregnant or lactating females Smokers (water pipe, cigar or cigarette smoking). Patients taking or have taken any drug that may cause gingival depigmentation as chloroquine, minocycline, zidovudine, chlorpromazine, ketoconazole and bleomycin .

Any cause for supplemental intake of vitamin C. Reported allergy to ascorbic acid or to any of its derivatives as reported in health questionnaire .

Clinically diagnosed periodontitis regarding the following criteria probing depth >3mm, clinical attachment loss ≥ 1mm and bleeding on probing > 10% .

Patients with poor oral hygiene, incompliant to treatment and persistence gingival inflammation after phase I periodontal therapy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Pigmentation scores | baseline (immediately before surgical depigmentation), one month, three months, six months, nine months and finally after 12 months post operatively
  Dummet oral pigmentation index (DOPI) ,score (0-3), 0 = pink tissue [no clinical pigmentation]; 1 = mild light brown tissue [mild clinical pigmentation]; 2 = medium brown or mixed brown and pink tissue [moderate clinical pigmentation]; or 3 = deep brown/ blue-black tissue (heavy clinical pigmentation)
Assessment of pigment surface area (SA) | baseline (immediately before surgical depigmentation), one month, three months, six months, nine months and finally after 12 months post operatively
  Standardized photos are taken and introduced into image J software after cropping interest area to calculate surface area of the pigment
Assessment of pigment intensity in terms of mean darkness value (MDV) | baseline (immediately before surgical depigmentation), one month, three months, six months, nine months and finally after 12 months post operatively
  Standardized photos are taken and introduced into image J software after cropping interest area to calculate intensity of pigment

SECONDARY OUTCOMES:
Patient satisfaction | After 12 months
  Satisfaction questionnaire Question Scoring
  Was the treatment painful?
  1. no pain; 2. Mild pain; 3. Severe pain
  Did you notice a cosmetic change 1 week after the treatment? 1. not at all; 2. moderate; 3. marked
  Did you notice a cosmetic change 6 week after the treatment?
  1. not at all; 2. moderate; 3. marked
  Did the treatment your expectations? 1. no; 2. yes; 3. Over and above
  Would you repeat the treatment if necessary?
  1. no; 2. yes; 3. Over and above
Histological response | baseline - 6 months -after a year
  Biopsies taken and stained with Fontana-Masson stain to calculate area fraction of the stained cells

CONTACTS AND LOCATIONS:
Overall Officials: Hala K. Abd-El-Gaber, Professor, Principal Investigator — Professor of Oral Medicine, Oral Diagnosis and Periodontology Faculty of Dentistry - Ain Shams University
Locations (1):
- Faculty AinShams University, Cairo, Egypt

REFERENCES:
- See also: Efficacy of surgical laser therapy in the management of oral pigmented lesions: A systematic review — http://pubmed.ncbi.nlm.nih.gov/28641206/
- See also: Gingival Depigmentation Using Scalpel Technique: A Case Report — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4374330/
- See also: An insight into gingival depigmentation techniques: The pros and cons — http://pubmed.ncbi.nlm.nih.gov/30202412/